CLINICAL TRIAL: NCT07327853
Title: Exploring the Prevalence and Potential Benefits of Fecal Immunochemical Test Before Ana After Use of Antiplatelet and Anticoagulant Agents
Brief Title: How Often Does the Fecal Test for Occult Blood Turn Positive After Using Blood Thinners?
Status: Not yet recruiting | Type: Observational
Sponsor: Jordan Collaborating Cardiology Group (Other)
Responsible Party: Sponsor
Other Study IDs: FIT/AP/AC#1.28.12.25
Record Dates: First submitted 2025-12-25; First posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Gastrointestinal Bleeding; Antiplatelet Agents; Oral Anticoagulant Therapy
Keywords: Occult fecal blood; Fecal Immunochemical Test (FIT); Gastrointestinal bleeding; Antiplatelet agents; Oral anticoagulant agents; Cardiovascular disease
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients to be prescribed oral antiplatelet and/or anticoagulant medications: The patients will have FIT performed before initiation of the oral antiplatelet and/or anticoagulant medications. Those with negative result will be followed up for 3 months after starting the medications and the FIT will be repeated. If the test turns positive, the patient will be referred for further evaluation be a gastroenterologist.
  Interventions: Diagnostic Test: Fecal Immunochemical Test (FIT)

INTERVENTIONS:
Diagnostic Test: Fecal Immunochemical Test (FIT) — A stool sample will be tested by the FIT test to examine the presence or absence of fecal occult blood. Each participant will be tested twice; one before starting the oral antiplatelet or anticoagulant agents and the second 3 months after the use of the medication.

SUMMARY:
Blood thinner medications used for cardiovascular disease can cause gastrointestinal bleeding. Early detection of invisible bleeding by performing occult fecal blood test (called fecal immunochemical test, or FIT) can uncover serious disease in the stomach and intestine and enable the treating physician to refer the patient for further evaluation.

DETAILED DESCRIPTION:
Oral anticoagulant and antiplatelet agents (AC/AP agents) are the cornerstone of treatment in patients with cardiovascular disease (CVD), including those with coronary artery disease, atrial fibrillation and deep vein thrombosis/pulmonary embolism. However, these agents are associated with risk of gastrointestinal (GI) bleeding. The bleeding can unmask certain GI pathologies early such as peptic ulcer disease, polyps and cancer. The fecal immunochemical test (FIT) is the most commonly used test utilized in clinical practice to detect occult fecal blood. There is scarcity of studies in the Middle East that evaluate the frequency of positive FIT in patients with CVD prescribed AC/AP agents with an initially negative FIT and who do not have history of bleeding or GI disease.

The concept of the study relies on performing FIT before AC/AP initiation, and if negative, the test will be repeated after 3 months. If the repeat test turns positive , these patients will be referred for further GI evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Have an indication to use oral antiplatelet or anticoagulant agent(s).
* Absence of past bleeding tendency of gastrointestinal disease.
* Agrees to have the test done (FIT).
* Agrees to sign the informed consent.

Exclusion Criteria:

* Presence of past bleeding tendency of gastrointestinal disease.
* Refusal to have the test done (FIT).
* Refusal to sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients to be included in the study are those who will be prescribed oral antiplatelet or anticoagulant (AP/AC) agents for a cardiovascular indication. They also should have no prior gastrointestinal disease. These patients will be evaluated over a period of 3 months after starting the AP/AC medication for the potential occurrence of occult gastrointestinal bleeding utilizing the fecal immunochemical test.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Positive Fecal Immunochemical Test | From the time of enrollment to the end of the study at 3 months
  A fecal specimen from each study participant will be tested for the presence or absence of fecal occult blood. This test will be performed before starting the oral antiplatelet or anticoagulant agents and will be repeated 3 months later.
Positive Fecal Immunochemical Test (FIT) | From enrollment to the end of the study at 3 months
  Positive Fecal Immunochemical Test (FIT) implies that the fecal sample obtained from each participant contains occult blood, denoting a bleeding source in the gastrointestinal system

CONTACTS AND LOCATIONS:
Locations (1):
- Istishari hospital, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Yes
The variables collected for each study participant will be provided upon request from the primary investigator including the baseline clinical features and lab results.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: April 2027 to December 2027